CLINICAL TRIAL: NCT03945084
Title: A Phase II, Randomized, Trial of Niraparib Versus Best Supportive Care as Maintenance Treatment In Patients With Locally Advanced Or Metastatic Urothelial Cancer Whose Disease Did Not Progress After First-line Platinum-based Chemotherapy
Brief Title: Maintenance With Niraparib In Patients With Advanced Urothelial Cancer After 1st-line Platinum-based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Principal Investigator, Massimo Di Maio, Associate Professor of Medical Oncology, Department of Oncology, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Meet-URO 12
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — niraparib

STUDY DESIGN:
Intervention Model Description: 2-arm, prospective, randomized (2:1 ratio), open-label, multi-centre, phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Arm (Experimental): Patients assigned to experimental arm will receive Niraparib 300 mg or 200 mg daily (based on weight and platelet count) plus best supportive care (BSC), in 28-day cycles, until disease progression or unacceptable toxicity or death.
  Interventions: Drug: Niraparib; Other: Best supportive care
- Control Arm (Other): Patients assigned to control arm will receive best supportive care alone, until disease progression or death.
  Interventions: Other: Best supportive care

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered as a flat-fixed, continuous daily dose:
  ≥77 kg and ≥150,000 µL: 300 mg (3 X 100 mg capsules) daily <77 kg or <150,000 µL: 200 mg (2 X 100 mg capsules) daily*
  * For patients whose starting dose is 2 capsules once daily, escalation to 3 capsules once daily will be permitted if no treatment interruption or discontinuation will be required during the first 2 cycles of therapy
  Other Names: Zejula
  Arms: Experimental Arm
Other: Best supportive care — In both treatment arms, Best Supportive Care (BSC) is defined as a comprehensive assessment of symptoms, with timely application of symptom control measures, in order to maximize patient's quality of life.
  BSC does not include any active antitumoral treatment, and will be given according to local guidelines and the normal practice of each participating institution.
  BSC will include use of opioid analgesics, other supportive drugs, radiotherapy, administered with the exclusive aim of improving tumor symptoms (e.g. pain, haematuria, etc.), according to Investigator's judgment.

SUMMARY:
This is a 2-arm, prospective, randomized (2:1 ratio), open-label, multi-centre, phase II study conducted in patients affected by unresectable, locally advanced or metastatic urothelial cancer receiving niraparib plus best supportive care versus best supportive care as maintenance therapy after a first-line platinum-based chemotherapy.

The primary objective of the trial is to evaluate the efficacy of niraparib plus Best Supportive Care (BSC) vs. BSC alone, as maintenance treatment, in terms of prolongation of progression-free survival (PFS), in patients with locally advanced or metastatic urothelial cancer that obtained disease control (objective response or stable disease) with first-line platinum-based chemotherapy.

DETAILED DESCRIPTION:
This is a 2-arm, prospective, randomized (2:1 ratio), open-label, multi-centre, phase II study conducted in patients affected by unresectable, locally advanced or metastatic urothelial cancer receiving niraparib plus best supportive care versus best supportive care as maintenance therapy after a first-line platinum-based chemotherapy.

The primary objective of the trial is to evaluate the efficacy of niraparib plus Best Supportive Care (BSC) vs. BSC alone, as maintenance treatment, in terms of prolongation of progression-free survival (PFS), in patients with locally advanced or metastatic urothelial cancer that obtained disease control (objective response or stable disease) with first-line platinum-based chemotherapy.

Poly-adenosine diphosphate ribose polymerase (PARP) inhibitors sensitivity is based on the presence of truncating and missense mutations in genes associated with the homologous recombination pathways. In The Cancer Genome Atlas dataset approximately 34% of bladder urothelial carcinoma harbored these mutations. Furthermore, in this study we plan to select a population potentially sensible to niraparib, by enrolling patients responding to platinum, indeed we know that there is a cross-sensitivity and a cross-resistance between platinum drugs and PARP inhibitors in urothelial carcinoma.

PFS is commonly adopted as primary endpoint in randomized phase II trials. Randomized design for phase II trials has been increasingly adopted in recent years, to allow a formal comparison between experimental and standard treatment. This should lead to a better interpretation of the results obtained with the experimental treatment, that are in most cases difficult to interpret in the absence of controls.

The sample size of the study is calculated with "relaxed" statistical criteria. The study design will verify if the experimental treatment (Niraparib) is promising enough to warrant a phase 3 trial for efficacy compared to observation.

A total of 65 PFS events are needed to provide 80% power to detect an hazard ratio (HR) of 0.57 (1.75), corresponding to a median increase in progression-free survival from 4 to 7 months, with one-tailed alpha 0.1.

With an accrual duration of 24 months, and additional 6 months of follow up after the completion of recruitment, 77 patient need to be randomized (26 assigned to control arm and 51 assigned to experimental arm) to obtain the 65 events needed.

Sample size of the phase II trial is too small to plan a formal analysis of interaction of treatment efficacy with type of response at first line treatment (i.e. objective response vs. stable disease). However, type of response to first line treatment will be among stratification factor for randomization, so the 2 treatment groups will be balanced. Exploratory subgroup analysis of treatment efficacy in patient who have obtained objective response with first line and in patients who have obtained stable disease with first line will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have histologically/cytologically confirmed, unresectable locally advanced or metastatic transitional cell carcinoma of the urothelium (transitional cell carcinoma either pure or mixed histology)
2. Measurable disease (per RECIST v1.1) prior to the start of first-line chemotherapy
3. Prior first-line chemotherapy must have consisted of at least 4 cycles and no more than 6 cycles of platinum containing regimen (cisplatin or carboplatin)
4. No evidence of progressive disease following completion of first-line chemotherapy (i.e., ongoing complete response (CR), partial response (PR), or stable disease (SD) per RECIST v1.1 guidelines )
5. Patients must be enrolled within 4 weeks of scans demonstrating stable disease/partial-complete response and no more than 6 weeks after receiving the last standard chemotherapy dose
6. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
7. Participant must be ≥ 18 years of age
8. Participant must have adequate bone marrow and organ function, defined as follows:

   * Absolute neutrophil count ≥ 1,500/µL
   * Platelets ≥ 100,000/µL
   * Hemoglobin ≥ 9 g/dL
   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
   * Total bilirubin ≤ 1.5 x ULN (≤2.0 in patients with known Gilberts syndrome) OR direct bilirubin ≤ 1 x ULN
   * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
9. Participant receiving corticosteroids is eligible if their dose is stable for least 4 weeks prior to initiating protocol therapy.
10. Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
11. Female participant has a negative urine or serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of non-childbearing potential. Non-childbearing potential is defined as follows (by other than medical reasons):

    * ≥45 years of age and has not had menses for >1 year
    * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
    * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment.

    Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
12. Participant must agree to not breastfeed during the study or for 180 days after the last dose of study treatment.
13. Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 180 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
14. Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent
15. Blood sample availability, to determine germline BRCA mutation status
16. Archived tumor tissue sample availability to determine homologous recombination deficiency (HRD) status

Exclusion Criteria:

1. Participant must not be simultaneously enrolled in any interventional clinical trial
2. Participant must not have had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
3. Participant must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
4. Participant must not have received radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
5. Participant must not have a known hypersensitivity to niraparib components or excipients.
6. Participant must not have been treated previously with a known PARP inhibitor agent
7. Participant must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
8. Participant must not have received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
9. Participant must not have experienced any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks.
10. Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
11. Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
12. Participant must not have a diagnosis of any other malignancy within 2 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast or of the cervix, low grade prostate cancer on surveillance without any plans for treatment intervention, or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease or symptoms.
13. Participant must not have history of or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan. However treated, stable and asymptomatic brain metastases are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
  PFS is defined as the time from the date of randomization to the earlier date of assessment of progression, or death by any cause in the absence of progression. Progression will be assessed following Response Evaluation Criteria In Solid Tumors (RECIST) criteria ( v.1.1 ), using investigator's review.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the percentage of patients with complete response (CR) or partial response (PR), as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (v.1.1)
Duration of response (DoR) | Up to 3 years
  DoR is defined as the time between the date of documented response and the date of first documented sign of clinical or radiological progression
Overall survival (OS) | Up to 3 years
  OS is defined as the time from the date of randomization to the date of death by any cause
Progression-free survival at 6 months | 6 months
  Progression-free survival at 6 month is defined as the rate of patients who are progression-free 6 months after randomization
Treatment-emergent adverse events (TEAEs) | Up to 3 years
  The study will collect information about the incidence of treatment-emergent AEs (TEAEs), coded and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Health-related quality of life | Up to 3 years
  The study will collect information about patient health-related quality of life using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. Multi-item scales are computed by calculating the mean raw scores of single items and transforming them linearly so that all scales range from 0 to 100. For single items, only linear transformation is performed. For functioning scales (i.e. those exploring physical, role, emotional, cognitive and social functioning and global health status), the higher the value the better the level of function; for symptoms scales and items, the higher the value the worse the severity of symptoms.

OTHER OUTCOMES:
BReast CAncer gene (BRCA) mutation status (exploratory) | Assessed on blood sample collected at baseline
  The study will collect blood sample from archival material of each patient at screening to assess BRCA mutation status.
Homologous Recombination Deficiency (HRD) status (exploratory) | Assessed on tumor tissue collected at baseline
  The study will collect tumor tissue from archival material of each patient at screening to assess HRD status

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Di Maio, MD, Principal Investigator — Department of Oncology, University of Turin
Locations (20):
- Italy (20):
  - Azienda Sanitaria Locale CN2 - Alba e Bra, Alba
  - Azienda USL Toscana Sud Est, Ospedale San Donato, Arezzo
  - Istituto Tumori Giovanni Paolo II - IRCCS, Bari
  - Presidio Ospedaliero Senatore A.Perrino, Brindisi
  - Azienda Ospedaliero-Universitaria, Cagliari
  - Azienda Ospedaliera Cannizzaro, Catania
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori IRCCS, Meldola
  - Istituto Nazionale Tumori IRCCS, Milan
  - Istituto Nazionale Tumori - Fondazione G.Pascale IRCCS, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - ASL Piacenza, Dipartimento Oncologico, Piacenza
  - Azienda Ospedaliero-Universitaria Pisana, Ospedale Santa Chiara, Pisa
  - Ausl - Irccs, Reggio Emilia
  - Irccs Crob, Rionero in Vulture
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Campus Biomedico, Roma
  - SCDU Oncologia Medica, AO Ordine Mauriziano, Torino
  - Presidio Ospedaliero Santa Chiara - APSS, Trento
  - AOU Santa Maria della Misericordia, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description of the results presented at ASCO GU 2022 — https://www.urotoday.com/conference-highlights/asco-gu-2022/asco-gu-2022-bladder-cancer/135451-asco-gu-2022-meet-uro12-phase-ii-study-of-niraparib-plus-best-supportive-care-vs-bsc-alone-as-maintenance-treatment-in-advanced-urothelial-carcinoma-patients-whose-disease-did-not-progress-after-first-line-platinum-based-chemotherapy.html